CLINICAL TRIAL: NCT06458634
Title: Impact of Weight Variation on Cop Displacement During Unperturbed Standing Conditions in Adolescents
Brief Title: Weight Variation on Cop
Status: Completed | Type: Observational
Sponsor: Amira Hussin Hussin Mohammed (Other)
Responsible Party: Sponsor-Investigator, Amira Hussin Hussin Mohammed, Associated professor, Delta University for Science and Technology
Organization: Delta University for Science and Technology (Other)
Other Study IDs: weight variation in COP
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Adolescent Overweight
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Underweight group: This group will be underweight group according to BMI- for age percentile growth chart ranged from BMI-for-age < 5th percentiles.
- Normal weight group: This group will be with normal weight according to BMI- for age percentile growth chart which ranged from BMI-for-age 5th to 85th percentiles
- Overweight group: This group will be an overweight group according to BMI- for age percentile growth chart which ranged from BMI-for-age 85th to 95th percentiles
- Obese group: This group will be obese group according to BMI- for age percentile growth chart which ranged from BMI-for-age > 95th percentiles and <99th percentile

SUMMARY:
This study will be conducted to investigate the impact of variant weights in adolescents during unperturbed standing conditions.

DETAILED DESCRIPTION:
200 adolescents from both sexes will be assigned to this study. They will be selected randomly from a secondary school student and first level university students. They will be assigned into four group of equal numbers according to (BMI) body mass index for age percentile obese group (n=50), overweight group (n=50), underweight group (n=50) and normal group weight (n=50).The FREEMED platform and FREESTEP software were used to assess the following parameters for each subject:

1. Sway length (mm).
2. The Maximum (peak) Oscillation of COP.
3. The minimum Oscillation of COP.

ELIGIBILITY:
Inclusion criteria:

* Their age will be ranging from 16 to 18 years.
* The sample will be selected according to (BMI-for Age percentile) growth charts according to CDC (Centers for Disease Control and Prevention) (appendix-1) (NCHS, 2014)
* All participant will be free from any musculoskeletal deformities.
* All participant are free of peripheral neuropathic diseases.
* They have no visual or auditory or vestibular disorders.
* They will able to understand, follow and execute instructions included in the testing analysis procedures.

Exclusion criteria:

* All adolescent associated with any musculoskeletal deformities.
* All adolescent associated with any foot deformity.
* All adolescent had a previous foot orthopedic procedure.
* All adolescent has visual or auditory or vestibular disorder.
* All adolescent has peripheral neuropathy.
* Adolescent with morbid obesity BMI >99th for age percentile (Barlow, 2007).

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: They will be assigned into four group of equal numbers according to (BMI) body mass index for age percentile obese group (n=50), overweight group (n=50), underweight group (n=50) and normal group weight (n=50).
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Sway length (mm) | through study completion, an average of 6 months
  The force platform was positioned in the middle of the test-taking silent room. In the static standing trial, each participant had the freedom to converse with their partner at any moment, provided that companion was either sitting or stood in front of them at a distance of roughly two meters. The AP and ML direction COP will be investigated using the data collected during the trial's eighty seconds. Depending on which of the six test trials was being given, the participant was advised to stand quietly and unperturbed throughout the test procedure, with their eyes either open or closed.
The Maximum (peak) Oscillation of COP | through study completion, an average of 6 months
  The force platform was positioned in the middle of the test-taking silent room. In the static standing trial, each participant had the freedom to converse with their partner at any moment, provided that companion was either sitting or stood in front of them at a distance of roughly two meters. The AP and ML direction COP will be investigated using the data collected during the trial's eighty seconds. Depending on which of the six test trials was being given, the participant was advised to stand quietly and unperturbed throughout the test procedure, with their eyes either open or closed.
The minimum Oscillation of COP | through study completion, an average of 6 months
  The force platform was positioned in the middle of the test-taking silent room. In the static standing trial, each participant had the freedom to converse with their partner at any moment, provided that companion was either sitting or stood in front of them at a distance of roughly two meters. The AP and ML direction COP will be investigated using the data collected during the trial's eighty seconds. Depending on which of the six test trials was being given, the participant was advised to stand quietly and unperturbed throughout the test procedure, with their eyes either open or closed.

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No